CLINICAL TRIAL: NCT05251532
Title: The Efficacy of Distortion Taping on Balance, Performance, Gait, Spasticity and Quality of Life in Ankle Varus Deformity in Children With Cerebral Palsy
Brief Title: The Efficacy of Distortion Banding on Outcome Measures in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPKT2
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy; Kinesio taping
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Group (KTG) (Experimental): Distortion taping with Kinesio Tex will be applied to the patients in addition to conventional rehabilitation through a pediatric physiotherapist.
  Interventions: Other: Kinesio Taping
- Conventional Rehabilitation Group (CRG) (Active Comparator): Conventional rehabilitation program will be applied to the patients through a pediatric physiotherapist.
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Kinesio Taping — In addition to Kinesio Tex tape distortion taping, conventional rehabilitation is applied.
  Arms: Kinesio Taping Group (KTG)
Other: Conventional Rehabilitation — Conventional rehabilitation practices are carried out
  Arms: Conventional Rehabilitation Group (CRG)

SUMMARY:
The aim of the study is to compare the conventional rehabilitation program and the distortion taping applied with Kinesio Tex tape in addition to conventional rehabilitation in children with hemiplegic or monoplegic cerebral palsy with ankle varus deformity.

DETAILED DESCRIPTION:
Conventional rehabilitation practices will be applied to the control group. In addition to Kinesio Tex tape distortion taping, conventional rehabilitation will be applied to the intervention group. It is aimed to evaluate the patients' balance, quality of life, performance test, spasticity level and gait quality.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy aged 4-12 years with unilateral involvement who are hemiplegic or monoplegic
* Cases with Gross Motor Function Classification (GMFCS) level 1 or 2
* Understanding simple commands and signing the consent form

Exclusion Criteria:

* Presence of equinus deformity
* Situations that may prevent assessments or communication
* Lack of cooperation during work
* Presence of surgery that may affect assessments, such as joint freezing
* Presence of botulinum toxin administration in the last 6 months
* Development of an allergic reaction on the skin to the tape

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
TUG | Change from Baseline TUG at 3 days
  Patients are asked to get up from a standard chair, walk 3 meters at a safe and comfortable pace, and return without stopping to sit back in the chair safely. The elapsed time is calculated. There is no score range in TUG.
SLS | Change from Baseline SLS at 3 days
  The one-leg standing test measures the time one is able to stand on one lower limb without support. There is no score range in SLS.
Modified Ashworth Scale (MAS) | Change from Baseline MAS at 3 days
  The Modified Ashworth Scale is a 6-point rating scale for gauging muscle resistance to passive movement. MAS is scored from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity.
WGS | Change from Baseline WGS at 3 days
  The scale allows for a multifactorial gait analysis, takes in to account 14 observable gait parameters divided into four sub-scales referring to particular phases of gait, i.e. stance phase, toe off, swing phase, andheel strike. WGS is scored from 13.35 to 42.0. Higher scores indicate higher impairment.
CHQ | Change from Baseline CHQ at 3 days
  The CHQ is a validated multidimensional instrument that measures the functional health and well-being of children and young people. CHQ is scored from 0 to 100. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet İmerci, PhD, Principal Investigator — Muğla Sıtkı Koçman University; İsmet Tümtürk, BSc, Principal Investigator — Ege University
Locations (1):
- Fethiye Private Son Atılım Special Education and Rehabilitation Center, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No